CLINICAL TRIAL: NCT00843258
Title: Immediate Treatment Compared With Active Sonographic Surveillance in the Management of Mild Hip Dysplasia in Newborn Infants: A Randomized, Controlled Trial
Brief Title: Treatment for Mild Hip Dysplasia in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: University of Bergen, Institute of SUrgical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mild hip dysplasia
Record Dates: First submitted 2009-02-11; First posted 2009-02-13 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Developmental Dysplasia of the Hip
Keywords: therapy; ultrasound; mild dysplasia
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Sonographic surveillance (No Intervention): Follow-up at 1.5 and 3 months (Ultrasound,Clinical examination), at 6 and 12 months (clinical examination, pelvic X-ray)
- Abduction treatment (Experimental): Treatment (abduction splint) from 0-6 weeks, follow-up at 1.5 and 3 months (clinical examination and ultrasound) and at 6 and 12 months (clinical examination and pelvic x-ray)
  Interventions: Device: Abduction treatment

INTERVENTIONS:
Device: Abduction treatment — Abduction treatment with a Frejka's pillow for 6 weeks
  Other Names: Pavlik harness
  Arms: Abduction treatment

SUMMARY:
Developmental dysplasia of the hip is the most common musculoskeletal disorder in infancy, with a reported prevalence of 2% of all newborns. Although newborn screening programs based on clinical examination with Ortolani and Barlow tests were introduced in the 1950's and 1960's with early abduction splinting of the 2% testing positive, the prevalence of late cases warranting surgery has remained stable, around one per 1000. This has led to the introduction of ultrasound as an additional diagnostic tool, resulting in treatment rates of until 5-6%. This three fold increase in abduction splinting treatment is partly due to the initiation of treatment of infants in whom mild hip dysplasia but no hip instability has been identified. The benefit of early treatment of mild dysplasia in a hip that is neither dislocated nor dislocatable is unclear. Further, abduction splinting is not without risk, with avascular necrosis being reported in around 1%. The investigators conducted a masked, randomized, controlled trial to examine whether mildly dysplastic but stable or instable hips would benefit from early treatment, as compared to watchful waiting.

DETAILED DESCRIPTION:
140 newborns with stable (not dislocatable or dislocated) but mildly dysplastic hips, born at the Maternity Hospital, Haukeland University Hospital, from 1997 onwards.

The newborns will be randomly assigned to one of two groups (number in sealed envelope, see flow chart). Because the newborns are recruited from a high risk group (60% with a positive family history and 35% breech), these risk factors are considered to be equally distributed in the two study groups. Stratification is therefore considered unnecessary.

For the controls, treatment will be started at age 1.5 months in cases of persistent dysplasia, i.e. a α-angle <50º, while treatment will be continued in the treatment group if the α-angle is ≤53º. At 3 months, treatment will be discontinued if the α-angle is ≥55º or started if α-angle is<55º. Treatment continued beyond 3 months will be discontinued when the AI is within two standard deviations according to the reference values from Tönnis and Brunken.

The study will require randomisation of 128 subjects into two equally sized groups to obtain 80% statistical power to detect a 3º difference of the α-angle. Less than 128 infants will be required to detect a similar difference in AI on radiography. To compensate for an expected rate of ineligibility and loss to follow-up of up to ten per cent, 140 patients will be enrolled.

PRACTICAL ISSUES The clinical hip-examinations will be performed at the maternity ward during day 1-3, by a physician with at least 2 years of pediatric experience. The hip joints will be classified as stable, unstable, dislocatable or dislocated. TM has the responsibility for the clinical re-examination prior to enrollement.

Ultrasound screening of newborns with increased risk for CDH is common practice at the maternity unit. Newborns eligible for the present study will be recruited from this high-risk group (about 13% of all newborns). To avoid inter-examination bias, all the ultrasound examinations will be performed by one examiner (KR), using a GE RT 3000, 5 MHz linear probe at KKB, and an ATL HDI 3000 machine with a 5 MHz linear probe or an Acuson 10XP, 5 MHz linear probe at the Section of Pediatric Radiology).

The ultrasound examinations will be performed according to a modified Graf procedure (Rosendahl), including both hip morphology and hip stability. Newborns with stable hips and a confirmed mild dysplasia on the second ultrasound examination will be re-examined clinically by TM, HR or TA prior to invitation to the study. After written informed consent has been given, the patient will attend the out patient clinic at BKB. A nurse will open the sealed envelope with a random number, and the newborn will enter the control or the treatment group. All data will be exported into SPSS by KR. RTL is the statistical adviser.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight > 2500 g
* Mild hip dysplasia on ultrasound day 1-2
* Written informed consent given

Exclusion Criteria:

* Birth weight less than 2500 g and/or severe congenital malformation(s)

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 1998-02; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
The acetabular index (AI), assessed from anterior-posterior pelvic radiographs obtained according to a standardized protocol at age 12 months | 12 months

SECONDARY OUTCOMES:
We also report the proportion of children requiring treatment in the first year of life and its duration, and the proportion of children in each group with radiological ossification delay or dysplasia at one year of age. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Rosendahl, PhD, Principal Investigator — Institute of Surgical Sciences, University of Bergen

REFERENCES:
- [Derived] Dwan K, Kirkham J, Paton RW, Morley E, Newton AW, Perry DC. Splinting for the non-operative management of developmental dysplasia of the hip (DDH) in children under six months of age. Cochrane Database Syst Rev. 2022 Oct 10;10(10):CD012717. doi: 10.1002/14651858.CD012717.pub2. PMID 36214650
- [Derived] Bruras KR, Aukland SM, Markestad T, Sera F, Dezateux C, Rosendahl K. Newborns with sonographically dysplastic and potentially unstable hips: 6-year follow-up of an RCT. Pediatrics. 2011 Mar;127(3):e661-6. doi: 10.1542/peds.2010-2572. Epub 2011 Feb 14. PMID 21321039
- [Derived] Rosendahl K, Dezateux C, Fosse KR, Aase H, Aukland SM, Reigstad H, Alsaker T, Moster D, Lie RT, Markestad T. Immediate treatment versus sonographic surveillance for mild hip dysplasia in newborns. Pediatrics. 2010 Jan;125(1):e9-16. doi: 10.1542/peds.2009-0357. Epub 2009 Dec 21. PMID 20026501